CLINICAL TRIAL: NCT01278225
Title: Effects of Neurofeedback on Neural Function, Neuromodulation, and Chemotherapy-Induced Neuropathic Pain
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-0675; NCI-2014-02452 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pain; Peripheral Neuropathy
Keywords: Neurofeedback; Neural Function; Neuromodulation; Chemotherapy-Induced Neuropathic Pain; Electroencephalogram; EEG; Biofeedback; BF; Quality of Life; QOL; Pain Quality Assessment Scale; PQAS; Brief Symptom Inventory; BSI; Sleep Disturbances; Fatigue; Questionnaires
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases; Parasomnias; Fatigue | interventions — Neurofeedback; Population Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EEG biofeedback (BF) Group: Group 1 will take part in a minimum of 2 neurofeedback training sessions each week for up to 10 weeks, for a total of up to 20 training sessions. After Group 1 completes neurofeedback training, both Groups to complete 10 questionnaires that were completed at baseline.
  Interventions: Behavioral: EEG biofeedback (BF) Group; Behavioral: Follow UP Questionnaires
- Wait-List Control (WLC) Group: Group 2 will be placed on a wait-list, will continue to receive standard care, will not take part in the neurofeedback training, but will take part in the follow-up visits. After Group 1 completes neurofeedback training, both Groups to complete 10 questionnaires that were completed at baseline.
  Interventions: Behavioral: Wait-List Control (WLC) Group; Behavioral: Follow UP Questionnaires

INTERVENTIONS:
Behavioral: EEG biofeedback (BF) Group — Group 1 will take part in a minimum of 2 neurofeedback training sessions each week for up to 10 weeks, for a total of up to 20 training sessions.
  Groups: EEG biofeedback (BF) Group
Behavioral: Wait-List Control (WLC) Group — Group 2 will be placed on a wait-list, will continue to receive standard care, will not take part in the neurofeedback training, but will take part in the follow-up visits.
  Groups: Wait-List Control (WLC) Group
Behavioral: Follow UP Questionnaires — After Group 1 completes neurofeedback training, both Groups to complete 10 questionnaires that were completed at baseline.

SUMMARY:
The goal of this study is to learn if using a non-invasive therapy called "neurofeedback training" can help teach patients ways to modify their own brain waves to decrease the perception of pain and improve quality of life.

DETAILED DESCRIPTION:
Baseline:

On Day 1, the following baseline tests and procedures will be performed:

* You will fill out 10 questionnaires about your pain, fatigue, how you have been feeling, and your general quality of life. The questionnaire packet may take up to 1 hour to complete.
* You will have an electroencephalograph (EEG -- a test that measures the electrical activity of the brain) performed. The EEG should take about 1 hour to complete.

Study Groups:

If you choose to take part in this study, after completing the baseline tests and procedures, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups.

Group 1 will take part in a minimum of 2 neurofeedback training sessions each week for up to 10 weeks, for a total of up to 20 training sessions. The neurofeedback training sessions may take place on any 2 days of the week and may be up to 5 times a week, if you are interested in training more quickly.

Group 2 will be placed on a wait-list, will continue to receive standard care, will not take part in the neurofeedback training, but will take part in the follow-up visits, described below. Group 2 will not take part in the neurofeedback training during Group 1's neurofeedback training period.

Neurofeedback Training (Group 1 only):

Neurofeedback training is a type of therapy that uses an EEG and a computer software program to measure brain wave activity. The neurofeedback training will be given in a video-game format and is designed to teach you ways to slowly re-train your brain wave activity by using "rewards" that you will hear and/or see when your brain waves change in the way the researchers are looking for.

With continuing feedback, coaching, and practice, researchers hope you will be able to learn how to produce the brain wave patterns that may help to reduce the perception of pain and improve quality of life.

For the EEG during each neurofeedback training session, researchers will place 1 or 2 electrodes on your scalp and 1 or 2 electrodes on each earlobe. The electrodes will measure and record your brain wave activity, similar to the way a doctor listens to your heart beat from the surface of your skin.

During each training session, you will sit quietly and relax while watching a computer screen. A neurotherapist will be present during each neurofeedback session to provide one-on-one assistance and guidance. Each neurofeedback training session will take up 1 hour to complete (about 15 minutes to get set up and about 45 minutes to complete the training session).

At each neurofeedback training session, the following tests and procedures will be performed:

* You will rate your pain on a scale of 0-10.
* You will be asked about any drugs you may be taking.

At the 10th training session only, you will also complete 3 questionnaires about your mood and pain. The questionnaires should take about 10 minutes to complete.

Follow-Up Visits (Both Groups):

If you are in Group 1:

* After you have completed neurofeedback training, and again 1 and 4 months later, you will fill out the same 10 questionnaires you completed at baseline.
* An EEG will be performed about 1 week after your last neurofeedback training session and again 4 months later.

If you are in Group 2:

* After Group 1 has completed neurofeedback training, and again 1 and 4 months later, you will fill out the same 10 questionnaires you completed at baseline.
* An EEG will be performed about 1 week after Group 1 has completed neurofeedback training (up to 10 weeks after baseline) and again 4 months later.

Length of Participation:

If you are in Group 1, after you complete the questionnaires at the follow-up visit 4 months after your last neurofeedback training session, your active participation on this study will be over.

If you are in Group 2, you will remain on study for up to 6 ½ months. If you choose to take part in the optional procedure, you will remain on study for up to 10 additional weeks to complete neurofeedback training.

This is an investigational study. The equipment used for neurofeedback training is FDA approved and commercially available equipment. Using neurofeedback equipment to teach patients ways to modify their own brain waves to decrease the perception of pain and improve quality of life is investigational.

Up to 80 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and read English, sign a written informed consent, and be willing to follow protocol requirements.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
3. Pain score >/= 4 on a 0-10 numeric pain scale and/or grade 3 neuropathic symptoms according to the National Cancer Institute's 4 point grading scale.
4. Pain must be related to chemotherapy (in the opinion of the treating physician).
5. Patients must have had neuropathic pain for a minimum of 3 months.
6. No plans to change pain medication regimen during the course of the study.
7. Off active chemotherapy treatment for minimum of 3 months.
8. Hormonal (e.g., tamoxifen or arimidex, etc.) and targeted (tarceva and avastin, etc.) therapies allowed as long as they will be continued during the course of the study.
9. Willing to come to MD Anderson for the therapy sessions; or willing to participate in the therapy sessions at their homes and live within a 45 minute drive of MDA main campus; or can participate in the therapy sessions from one of MDA's Regional Care Centers.

Exclusion Criteria:

1. Patients who are taking any antipsychotic medications.
2. Patients with active central nervous system (CNS) disease, such as clinically-evident metastases or leptomeningeal disease, dementia, or encephalopathy.
3. Patients who have ever been diagnosed with bipolar disorder or schizophrenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving chemotherapy at UT MD Anderson Cancer Center in Houston, Texas
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-02 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Effects of Individualized Electroencephalogram (EEG) Biofeedback Treatment Regimen on Perceptions of Chemotherapy-Induced Neuropathic Pain | 10 weeks
  After Group 1 has completed neurofeedback training, both Groups will fill out the same 10 questionnaires that were completed at baseline. An EEG will be performed on both Groups about 1 week after Group 1 completes last neurofeedback training, and again 4 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Prinsloo, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Prinsloo S, Novy D, Driver L, Lyle R, Ramondetta L, Eng C, Lopez G, Li Y, Cohen L. The Long-Term Impact of Neurofeedback on Symptom Burden and Interference in Patients With Chronic Chemotherapy-Induced Neuropathy: Analysis of a Randomized Controlled Trial. J Pain Symptom Manage. 2018 May;55(5):1276-1285. doi: 10.1016/j.jpainsymman.2018.01.010. Epub 2018 Feb 5. PMID 29421164
- See also: University of Texas MD Anderson Cancer Center Website — http://www.utmdanderson.org